CLINICAL TRIAL: NCT02302963
Title: Unified Safety System (USS) Virginia Closed-Loop Versus Sensor Augmented Pump Therapy for Hypoglycemia Reduction in Type 1 Diabetes
Brief Title: USS Virginia Closed-Loop Versus SAP Therapy for Hypoglycemia Reduction in T1D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other); TypeZero Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17725; 1DP3DK101055 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2014-11-27 (Estimated); Results first posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1 (T1DM); Diabetes Assistant (DiAs); Artificial Pancreas (AP) System; Closed-Loop Control (CLC); Unified Safety System (USS) Virginia; Sensor Augmented Pump (SAP); Low Blood Glucose Index (LBGI); Continuous Glucose Monitor (CGM); inControl Diabetes Management Platform
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP System (DiAs or inControl) with USS Virginia (Experimental): Subject will complete an 8-hour inpatient assessment of hypoglycemia counterregulation. Subject will then proceed through 7 weeks of training and use of the AP System with USS Virginia and study pump. The inpatient testing will be repeated after wearing the AP System at home.
  Interventions: Device: AP System (DiAs or inControl) with USS Virginia
- Sensor-Augmented Pump Therapy (Placebo Comparator): Subject will complete an 8-hour inpatient assessment of hypoglycemia counterregulation. Subject will then wear a continuous glucose monitor and their own insulin pump at home for 5 weeks. The inpatient testing will be repeated at the completion of the 5 weeks at home.
  Interventions: Device: Sensor-Augmented Pump Therapy (placebo)

INTERVENTIONS:
Device: AP System (DiAs or inControl) with USS Virginia — Subject will participate in two 24-hour study insulin pump and AP System training sessions. At the conclusion of each training session, subject will wear the equipment at home for a total of 5 weeks.
  Arms: AP System (DiAs or inControl) with USS Virginia
Device: Sensor-Augmented Pump Therapy (placebo) — Subject will participate in 5 weeks use of CGM and personal insulin pump at home.
  Arms: Sensor-Augmented Pump Therapy

SUMMARY:
This is a randomized, controlled trial of Unified Safety System (USS) Virginia closed-loop versus sensor-augmented pump (SAP) therapy for hypoglycemia prevention in subjects with type 1 diabetes and hypoglycemia unawareness and/or risk for hypoglycemia.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of the control system in reducing hypoglycemia by comparing, in a randomized study, 24 hour control with USS Virginia versus sensor augmented pump (SAP) therapy in subjects with type 1 diabetes and hypoglycemia unawareness and/or risk for hypoglycemia. We will also evaluate the effectiveness of the control system to improve hypoglycemia counterregulation, hypoglycemia awareness, and overall glycemic control. To achieve this goal, we will conduct pre- and post-intervention inpatient assessments of hypoglycemia counterregulation and symptom awareness. Subjects randomized to USS Virginia will participate in two training visits at a monitored outpatient setting for the step-wise deployment of the cell phone based Artificial Pancreas (AP) System at home. The first training visit includes training on the study pump and AP System followed by 1 week use of AP System at home in Pump mode. The second training visit includes additional training on USS Virginia+AP System and confirmation of independent use by the subject followed by 4 week use of the AP System at home in Closed Loop mode. Subjects randomized to sensor-augmented pump therapy will complete 5 weeks of CGM with the home pump.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of type 1 diabetes for at least 1 year. For an individual to be enrolled at least one criterion from each list must be met:

Criteria for documented hyperglycemia (at least 1 must be met):

1. Fasting glucose ≥126 mg/dL (confirmed)
2. Two-hour oral glucose tolerance test (OGTT) glucose ≥200 mg/dL (confirmed)
3. HbA1c ≥6.5% (confirmed)
4. Random glucose ≥200 mg/dL with symptoms
5. No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes or in the opinion of the investigator participant has history consistent with type 1 diabetes.

Criteria for requiring insulin at diagnosis (at least 1 must be met):

1. Participant required insulin at diagnosis and continually thereafter
2. Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
3. Participant required insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually thereafter

   * Use of insulin for the last 12 months or more
   * Use of an insulin infusion pump for the last 6 months or longer
   * Age 12-70 years old
   * HbA1c <10.0% as measured with DCA2000 or equivalent device; if HbA1c <6.0% then total daily insulin must be ≥0.5 U/kg
   * Risk of hypoglycemia or hypoglycemia unawareness as defined by any of the following:
   * Clarke Hypoglycemia Perception Awareness questionnaire score of ≥4.
   * Average Daily Risk Range (ADRR) >40 as assessed from Self-Monitoring Blood Glucose (SMBG) readings from the prior month. Subject must have a glucometer that can be downloaded for this assessment. The subjects may alternatively provide a spreadsheet of their past 30 days of blood glucose values.
   * Low Blood Glucose Index (LBGI) >2.5 as assessed from SMBG from the prior month or LBGI >1.1 as assessed from 1 week of CGM readings from the prior three weeks. Subject must have a glucometer or CGM that can be downloaded for this assessment. For the glucometer data, the subjects may alternatively provide a spreadsheet of their past 30 days of blood glucose values.
   * Subject reports no recognition of hypoglycemia until the glucose is <60 mg/dL and no adrenergic symptoms at glucose of 60 mg/dL (shakiness, palpitations, diaphoresis).
   * Able to speak and read English and use basic technology such as a cell phone.
   * Currently using an insulin-to-carbohydrate ratio to calculate meal bolus sizes.
   * Access to Internet or cell phone service in the subject's local environment.
   * Willingness to maintain uninterrupted availability via personal cell phone at all times during the study.
   * Willingness to perform SMBG testing 4-6 times daily (before meals, about 2 hours after meals and at bedtime, before driving, before exercise, and as indicated) during the interventional phases of the study.
   * Living with a diabetes care partner ≥18 years old who meets the following inclusion criteria:
   * Committed to potentially (if randomized to DiAs) participating in all training activities involving DiAs components and emergency procedures,
   * Knowledgeable at all times of the participant's location during the day when closed loop is in use,
   * Committed to maintaining uninterrupted availability via personal cell phone,
   * Being present and available to provide assistance when the closed loop system is being used at night,
   * Able to speak and read English and use basic technology such as a cell phone, and
   * Absence of known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:
   * Inpatient psychiatric treatment in the past 6 months,
   * Current or recent abuse of alcohol or recreational drugs by history
   * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication, or disease in the judgment of the investigator will affect the completion of the protocol.

Exclusion Criteria:

The presence of any of the following is an exclusion for the study:

1. Admission for diabetic ketoacidosis in the 12 months prior to enrollment.
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 3 months prior to enrollment.
3. Hematocrit less that the lower limit of normal for the assay.
4. Pregnancy, breast-feeding, or intention of becoming pregnant over time of study procedures; If female and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative urine pregnancy test will be required for all premenopausal women who are not surgically sterile. Subjects who become pregnant will be discontinued from the study.
5. Conditions which may increase the risk of induced hypoglycemia such as: known coronary artery disease, congestive heart failure, history of any cardiac arrhythmia (benign premature atrial contractions and premature ventricular contractions allowed), history of seizure disorder, history of cerebrovascular event or transient ischemic attack, hypoglycemia-induced migraine within the last 6 months, or neurological disease.
6. Cystic fibrosis
7. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:
8. Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's diabetes care partner
9. Presence of a known adrenal disorder
10. Abnormal liver function tests (transaminase >3 times the upper limit of normal); testing required for subjects taking medications known to affect liver function or with diseases known to affect liver function
11. Abnormal renal function test results (estimated Glomerular filtration rate (GFR) <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
12. Active gastroparesis
13. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
14. Uncontrolled thyroid disease (TSH undetectable or >10 mIU/L); testing required within 3 months prior to admission for subjects with a goiter, positive antibodies, or who are on thyroid hormone replacement, and within one year otherwise
15. Current or recent abuse of alcohol or recreational drugs by patient history
16. Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis)
17. Any skin condition in the area of insertion that prevents safe sensor or pump placement (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
18. Diagnosed with celiac disease and not currently following a gluten free diet

    * A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication, or disease in the judgment of the investigator will affect the completion of the protocol
    * Current use of any of the following drugs and supplements:
19. Any medication being taken to lower blood glucose, such as Pramlintide, Metformin, Glucagon-like peptide-1 (GLP-1) Analogs such as Liraglutide, and nutraceuticals intended to lower blood glucose
20. Beta blockers
21. Oral glucocorticoids
22. Pseudoephedrine
23. Any other medication that the investigator believes is a contraindications to the subject's participation

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacey M. Anderson, MD, Principal Investigator — UVA Center for Diabetes Technology; Bruce Buckingham, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NIH's Data Sharing Policy on sharing research resources for research purposes to the scientific community will be followed. Data will be stored in a Data Archive Database includes CGM-insulin delivery time series, meal content, boluses, & exercise will be deidentified & retrievable only by subject ID number. The data's real value lies in their precise time stamps - each reading is coded by date & time which makes possible the data to be related to the subjects' daily routine. Individual patterns of demographic & insulin treatment parameters leave open a remote possibility of deductive disclosure of subjects with unusual characteristics. Data can be made available only under a Data-Sharing Agreement that includes: (1) a commitment to using the data only for research purposes & not to identify participants; (2) a commitment to securing the data using appropriate computer technology; & (3) a commitment to destroying or returning the data after analyses are completed.
Supporting Information: Study Protocol, ICF
Time Frame: After publication of the primary manuscript, published in Diabetes Technology and Therapeutics, Volume 21, Number 6, 2019
Access Criteria: Study outcomes are presented in the primary manuscript. Raw data can be shared via data sharing agreement, as described in the Data Sharing Plan.

REFERENCES:
- [Result] Anderson SM, Buckingham BA, Breton MD, Robic JL, Barnett CL, Wakeman CA, Oliveri MC, Brown SA, Ly TT, Clinton PK, Hsu LJ, Kingman RS, Norlander LM, Loebner SE, Reuschel-DiVirglio S, Kovatchev BP. Hybrid Closed-Loop Control Is Safe and Effective for People with Type 1 Diabetes Who Are at Moderate to High Risk for Hypoglycemia. Diabetes Technol Ther. 2019 Jun;21(6):356-363. doi: 10.1089/dia.2019.0018. Epub 2019 May 16. PMID 31095423

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 85 subjects consented; 20 didn't meet eligibility criteria & 21 subjects withdrew/dropped (18 prerandomization, 1 control, 2 exp). Reasons for withdrawal included scheduling conflicts (5), travel cost (1), interest in a different CLC trial (2), dislike of DiAs (1), alarm fatigue (1), steroid injection (1), and loss communication (10). 44 subjects completed. CGM data missing for 2 of the 44 subjects (1 control, 1 exp); therefore, 42 subjects included in final analysis.
Pre-assignment Details: After study eligibility was met, subjects completed 1 week of baseline blinded CGM and SMBG at least four times daily. If LBGI >1.1 was confirmed by blinded CGM, the subject was randomized to USS Virginia AP experimental treatment or sensor-augmented pump control treatment.
Period: Overall Study
Arm/Group | AP System (DiAs or inControl) With USS Virginia | Sensor-Augmented Pump Therapy
Started | 25 | 24
Completed | 22 | 22
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Steroid injection | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AP System (DiAs or inControl) With USS Virginia | Sensor-Augmented Pump Therapy | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (3.3) | 38.0 (3.3) | 38.2 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 22 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hypoglycemia During Closed Loop Control (Assessed by Low Blood Glucose Index [LBGI])
Description: Change in hypoglycemia during the study on USS Virginia versus Sensor Augmented Pump (SAP) as assessed by Low Blood Glucose Index (LBGI) from Continuous Glucose Monitoring (CGM) during 1 week of baseline blinded use versus during the last week of intervention. The LBGI is a metric of the frequency and severity of hypoglycemia, based on an increasing weighting of progressively low glucose readings. The LBGI will be higher for someone with a higher percentage of low blood glucose readings or more extreme hypoglycemic episodes. Reference: Kovatchev BP. Metrics for Glycaemic Control: from HbA1c to Continuous Glucose Monitoring. Nature Reviews Endocrinology 2017; 13: 425-436. PMID: 28304392
Time Frame: 2 weeks total: one week of baseline blinded use to compute LBGI-Pre versus use during the last week of intervention to compute LBGI-Post
Measure: Mean (Standard Deviation); unit: low blood glucose index
Arm/Group | AP System (DiAs or inControl) With USS Virginia | Sensor-Augmented Pump Therapy
Number analyzed (Participants) | 21 | 21
low blood glucose index
  LBGI (after 1 week of blinded CGM) | 2.51 (1.17) | 2.1 (1.05)
  LBGI (last week of intervention after 5 weeks of study participation) | 1.28 (0.5) | 1.79 (0.98)
Statistical Analysis 1: Comparison: AP System (DiAs or inControl) With USS Virginia vs Sensor-Augmented Pump Therapy; Test type: Other — Analysis of Variance; p < 0.001, GLM Repeated Measures; Repeated-measures general linear model was used to compare HCLC versus SAP data. A P-value of < 0.001 was considered the threshold for significance

ADVERSE EVENTS:
Time Frame: Up to 14 weeks of study participation (visit 2 through visit 6)
Arm/Group | AP System (DiAs or inControl) With USS Virginia | Sensor-Augmented Pump Therapy
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 8/22 | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AP System (DiAs or inControl) With USS Virginia (N=22) | Sensor-Augmented Pump Therapy (N=22)
Moderate hyperglycemia, mild ketonemia (Endocrine disorders) | 1 (1) | 0 (0)
Moderate hyperglycemia, moderate ketonemia (Endocrine disorders) | 3 (3) | 2 (2)
Mild ketonemia (Endocrine disorders) | 2 (2) | 0 (0)
Soccer injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Respiratory illness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
IV Site Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Arm fracture from fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — outpatient surgery for spiral fracture of arm
Fever (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Vasovagal event (Nervous system disorders) | 1 (1) | 1 (2)

LIMITATIONS AND CAVEATS:
CGM data were missing for 2 of the 44 subjects (1 control and 1 experimental) and outcomes could not be reliably computed. Therefore, 42 subjects were included in the final analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02302963/Prot_SAP_000.pdf